CLINICAL TRIAL: NCT00772083
Title: Caring for Those Who Share: Improving the Health of Wisconsin Blood Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Healthier Wisconsin Partnership Program (Unknown); Versiti Blood Health (Other); National Anemia Action Council (Other)
Responsible Party: Kenneth G. Schellhase, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PRO00008944
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Anemia; Colorectal Cancer
MeSH Terms: conditions — Anemia; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Educational brochure
- 2 (Active Comparator): standard approach currently being used
  Interventions: Behavioral: Standard pamphlet

INTERVENTIONS:
Behavioral: Educational brochure — This brochure will educate anemic blood donors regarding the possible causes of their anemia, and based on age will make recommendations for who should seek consultation with a physician.
  Arms: 1
Behavioral: Standard pamphlet — The BloodCenter of Wisconsin's default action when a potential donor has been found to be anemic is to provide a standard pamphlet with very basic nutritional information.
  Arms: 2

SUMMARY:
Blood donors are a precious community resource. Each month at Blood Center of Wisconsin (BCW), 200 men and 600 women over age 50 are turned away ("deferred") because of anemia. In those over 50, anemia may signal serious underlying disease such as colorectal cancer (CRC). CRC is the #3 cause of cancer death in Wisconsin with more than 1,000 deaths in 2006. Yet with proper testing CRC outcomes can be improved by early diagnosis. This project will focus on a population of deferred older blood donors to develop and test educational materials that will motivate donors to seek medical attention for their anemia, so that the underlying cause is diagnosed and treated. This project has the potential to lead to better CRC outcomes in Wisconsin blood donors.

ELIGIBILITY:
Inclusion Criteria:

* adult blood donors who have been "deferred" (not allowed to donate) due to low blood count, specifically all male donors found to have hematocrit < 38% and to all female donors over 50 years old found to have hematocrit < 36%

Exclusion Criteria:

* deferred donors who have previously donated more than 3 times in the past year, as their anemia is more likely due to frequent donation
* women less than 50 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
self-reported seeking of medical care for diagnosis of anemia found at time of blood donation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G Schellhase, MD MPH, Principal Investigator — Medical College of Wisconsin; Alan Mast, MD PHD, Principal Investigator — Versiti Blood Health
Locations (1):
- BloodCenter of Wisconsin, Milwaukee, Wisconsin, United States